CLINICAL TRIAL: NCT04204174
Title: Identification of P-cresyl Sulfate Producer Phenotype by Oral Tyrosine Challenge Test: Interactions Among Diet, Gut Microbiota, and Host Genome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Ting-Yun Lin, Nephrologist, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08-X-108
Record Dates: First submitted 2019-12-08; First posted 2019-12-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Chronic Kidney Diseases; Healthy
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Tyrosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tyrosine loading (Experimental)
  Interventions: Dietary Supplement: Tyrosine, brand name: myprotein

INTERVENTIONS:
Dietary Supplement: Tyrosine, brand name: myprotein — tyrosine at a dose of 100 mg/kg is then administered orally to the participants once

SUMMARY:
Patients with chronic kidney disease (CKD) display a substantial increase in cardiovascular disease (CVD). Moreover, the prognosis of CVD in CKD is extremely poor. Understanding the pathophysiology of CVD in CKD might help to develop treatment strategies to reduce its morbidity and mortality. Compelling evidence suggests that the uremic milieu itself plays a critical role in the development and progression of CVD in CKD. The gut microbiota is markedly altered in CKD. Fermentation of protein and amino acids by certain gut microbiota results in the generation of different uremic toxins. p-cresyl sulfate (PCS) is among the most representative gut-derived uremic toxins implicated in the pathogenesis of CVD in CKD. However, there remained no clear cut-off value of fasting plasma PCS for unfavorable clinical outcomes.

Thus, we plan to establish an oral tyrosine challenge test (OTCT) integrated with dietary patterns, gut microbiome, and serum biochemistry to assess PCS synthesis capacity from host-diet-microbiota interactions.

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) display a substantial increase in cardiovascular disease (CVD). Moreover, the prognosis of CVD in CKD is extremely poor. Understanding the pathophysiology of CVD in CKD might help to develop treatment strategies to reduce its morbidity and mortality. Traditional CV risk factors for the general population, such as diabetes mellitus, high blood pressure, and dyslipidemia, are more common in patients with CKD, but cannot entirely explain the increased CV risk. Compelling evidence suggests that the uremic milieu itself plays a critical role in the development and progression of CVD in CKD. The gut microbiota is markedly altered in CKD. Fermentation of protein and amino acids by certain gut microbiota results in the generation of different uremic toxins. p-cresyl sulfate (PCS) is among the most representative gut-derived uremic toxins implicated in the pathogenesis of CVD in CKD (JAHA 6:e005022, 2017). However, there remained no clear cut-off value of fasting plasma PCS for unfavorable clinical outcomes (Clin J Am Soc Nephrol 4:1551-8, 2009). The benefit of adding an orally administered adsorbent (AST-120) to standard therapy in unselected patients with moderate to severe CKD is also not supported by data from a recent randomized controlled trial (J Am Soc Nephrol 26:1732-46, 2015).

It has been shown that uremic toxicity is related to the peak rather than the time-averaged urea concentration (Perit Dial Int 9:257-60, 1989). PCS is mainly produced from the metabolism of dietary tyrosine by gut bacteria. PCS concentration may fluctuate widely from time to time in response to meals. A postprandial plasma PCS might theoretically reflect the pathophysiological level of PCS. Thus, we plan to establish an oral tyrosine challenge test (OTCT) to simulate the postprandial plasma PCS among patients with CKD to identify "PCS producers" who are likely to be at high risk for CVD and are more likely to respond to adsorbent therapy. The OTCT survey is integrated with dietary patterns, gut microbiome, and serum biochemistry to assess PCS synthesis capacity from host-diet-microbiota interactions.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease stages 3-5D patients OR
* healthy volunteers

Exclusion Criteria:

* subjects who has ever exposure to antibiotics or probiotics within the 3 months before entering the study
* patients with active gastrointestinal diseases or recent gastrointestinal discomfort (such as abdominal pain or diarrhea)
* patients with liver cirrhosis
* pregnant or breastfeeding women

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
level of serum p-cresyl sulfate | the area under curve of serum p-cresyl sulfate
  serum p-cresyl sulfate level after oral tyrosine loading up to 48 hours

SECONDARY OUTCOMES:
level of serum phenyl sulfate | the area under curve of serum phenyl sulfate
  serum phenyl sulfate level after oral tyrosine loading up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Yun Lin, MD., Principal Investigator — Taichung Tzu Chi Hospital
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
We have decided yet.